CLINICAL TRIAL: NCT05921526
Title: Effectiveness of Point-of-care Lung Ultrasound vs Chest X-ray for the Management of Childhood Lower Respiratory Infections in Low-resource Setting: Single Center, Pragmatic, Open-label, Randomized, Controlled, Non-inferiority Clinical Trial
Brief Title: Effectiveness of Point-of-care Lung Ultrasound for the Management of Childhood Lower Respiratory Infections
Acronym: ELUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nagasaki University (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Siddhi Memorial Foundation (Other)
Responsible Party: Principal Investigator, Suraj BHATTARAI, PhD Fellow, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELUS study
Record Dates: First submitted 2023-05-18; First posted 2023-06-27 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-05

CONDITIONS: Lower Respiratory Infection; LRTI; Pneumonia; Bronchiolitis
Keywords: Point-Of-Care Lung UltraSound; POCLUS; Lung POCUS
MeSH Terms: conditions — Pneumonia; Bronchiolitis | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Point-of-care lung ultrasound
  Interventions: Diagnostic Test: Point-of-care lung ultrasound
- Control (Active Comparator): Chest X-ray
  Interventions: Diagnostic Test: Chest X-ray (digital images)

INTERVENTIONS:
Diagnostic Test: Point-of-care lung ultrasound — Participants assigned to the intervention group will receive POCLUS which will be performed by one of the trained pediatricians. The procedure involves 12 views: two anterior views, two lateral views and two posterior views on both chest walls
  Other Names: POCLUS
  Arms: Intervention
Diagnostic Test: Chest X-ray (digital images) — Participants assigned to the chest X--ray group will be sent to the Radiology department to get a CXR (digital) which will be performed by radio technicians like in routine care. Anteroposterior and/or posteroanterior chest images will be obtained. Reading/ reporting of the digital images will be done by both the radiologist and the enrolling pediatrician. The image/ clinical expert review panels (IERP/ CERP) will also have access to the images for review.
  Other Names: CXR
  Arms: Control

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of point-of-care lung ultrasound versus chest X-ray for the management of childhood lower respiratory infections in a low-resource setting.

The main question it aims to answer is:

Is point-of-care lung ultrasound as effective as chest X-ray for the management of childhood LRIs in a low-resource setting?

Participants will be assigned to either a point-of-care lung ultrasound group (intervention) or a chest X-ray group (control), to compare the effect on overall case management and various clinical outcomes (time to symptom resolution, rate of antibiotic use, length of stay, treatment costs).

DETAILED DESCRIPTION:
Background:

Lower respiratory infections (LRIs) are the leading causes of mortality in children of low-middle income countries (LMICs) including Nepal; pneumonia being the major killer in under-5 population. Often, the cause of mortality is the delay in diagnosis and treatment, particularly when clinical assessments do not hint toward a diagnosis. In resource-limited settings, routine availability of chest X-ray (CXR) service is a challenge, it can be hazardous to children due to exposure to ionizing radiation. The Point-Of-Care Lung UltraSound (POCLUS) could be an alternative solution for the diagnosis and management of LRIs. Studies have already shown that lung ultrasound has a higher sensitivity and specificity than CXR in diagnosing childhood LRIs, however, none of the studies have yet evaluated its role in overall case management.

Methods:

Prospective, single-center, pragmatic, open-label, randomized, controlled, non-inferiority clinical trial, which will be conducted in the outpatient and emergency departments of a pediatric hospital in Nepal. A total of 616 children with clinical suspicion of LRI and requiring chest imaging will be randomized at 1:1 allocation to the intervention (POCLUS) and control (CXR) arms. Pediatricians will be trained to perform lung ultrasonography in children.

Outcomes:

Primary outcome is the proportion of 'correctly (effectively) managed' cases. Secondary outcomes include the proportion of cases with 'change in diagnosis and management plan due to intervention', time to symptom resolution, rate of antibiotic use, length of stay, and in-hospital costs, compared between intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Children with a suspected lower respiratory infection (LRI) brought to the outpatient or emergency department,
* Requiring chest image for evaluation at baseline.

Exclusion Criteria:

* Children already hospitalized, received antibiotics, or had chest imaging at the hospital;
* Follow-up (treated within the past 4 weeks) or referred cases;
* Critical patients requiring emergency life-saving support including oxygen;
* Children with one or more danger signs (lethargy or loss of consciousness, convulsion, unable to eat or vomiting everything, cyanosis, excess irritability)

Ages: 2 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 616 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Correct management plan at the baseline on the basis of clinical assessment and chest image findings | From the date of randomization until the final disposition of patient (i.e. discharge, refer), assessed up to 3 weeks. In case of non-hospitalized participants, outcomes evaluated during 2nd follow up (day 7-10 of enrollment), assessed up to 2 weeks.
  Proportion of participants who are prescribed a correct management plan at the baseline on the basis of clinical assessment and chest image findings, either point-of-care lung ultrasound or chest X-ray

SECONDARY OUTCOMES:
Change in diagnosis and management plan | From the date of randomization until Day3-5 of enrollment, assessed up to 1 week.
  * Diagnosis and Management Plan 1: Enrolling physician will fill a case report form with initial diagnosis and management plan (plan 1) based on the clinical assessment and LUS/CXR findings at baseline.
  * Decision regarding actual diagnosis and management plan (1a) is on treating physician's discretion.
  * Diagnosis and Management Plan 2: Enrolling physician will fill a second case report form (exactly same to the first one) on Day3-5 of enrollment with the diagnosis and management plan based on clinical assessment, chest image(s), and lab investigations.
  This outcome is measured in hospitalized cases only.
Time to symptom/sign resolution | From the date of randomization until disposition (i.e. discharge, referral) or symptom resolution criteria is met, whichever is earlier, assessed up to 3 weeks.
  In hospitalized cases only
Length of stay at hospital | From the date of randomization until disposition (i.e. discharge, referral), assessed up to 3 weeks.
  In hospitalized cases only
Rate of antibiotic use | From the date of randomization until disposition (i.e. discharge, referral), assessed up to 3 weeks.
  In hospitalized cases only
In-hospital treatment costs | From the date of randomization until disposition (i.e. discharge, referral), assessed up to 3 weeks.
  In hospitalized cases only

CONTACTS AND LOCATIONS:
Overall Officials: Suraj Bhattarai, MBBS, MSc, DTM&H, Principal Investigator — LSHTM/Nagasaki U/Siddhi Memorial Hospital; Bhim Dhoubhadel, MBBS MTM PhD DipPaed DTM&H, Principal Investigator — Nagasaki University; Shunmay Yeung, PhD MBBS FRCPCH MRCP DTM&H, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Siddhi Memorial Hospital, Bhaktapur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, deidentified participant data, and study tools may be shared with other researchers upon reasonable request, and decided by the investigators.
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol will be published in a journal. Clinical study report may be shared after the study is closed.
Access Criteria: It will be decided by the team of principle investigators.